CLINICAL TRIAL: NCT02423447
Title: Comparison of the Airway Clearance Efficacy of Electro Flo 5000 and the G5 Flimm-Fighter in Patients With Cystic Fibrosis (CF)
Brief Title: Comparison of the Airway Clearance Efficacy of Electro Flo 5000 and the G5 Flimm-Fighter in Patients With CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Carlos Milla, Associate Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 27689
Record Dates: First submitted 2015-02-03; First posted 2015-04-22 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electro-Flo Arm (Active Comparator): The patients were randomized to a series of airway clearance sessions with Electro-Flo on Day 1 and G5 on Day 2.
  Interventions: Device: Electro-Flo Intervention
- G5 Arm (Active Comparator): The patients were randomized to a series of airway clearance sessions with G5 on Day 1 and Electro-Flo on Day 2.
  Interventions: Device: G5 Intervention

INTERVENTIONS:
Device: Electro-Flo Intervention — An assigned respiratory therapist performed airway clearance on each participant with the Electro-Flo device following the 2012 CFF therapy guidelines
  Arms: Electro-Flo Arm
Device: G5 Intervention — An assigned respiratory therapist performed airway clearance on each participant with the G5 device following the 2012 CFF therapy guidelines
  Arms: G5 Arm

SUMMARY:
It is the goal of the proposed study to compare the efficacy, as assessed primarily by sputum weight, of these two different devices (the Electroflo 500 and the G5 Flimm-Fighter) for airway clearance (AC) in CF patients with mild to moderate lung disease, who have stable lung health and perform AC at home as part of their routine therapeutic regimen.

DETAILED DESCRIPTION:
The investigators hope to enroll 25 patients with cystic fibrosis (with daily sputum production) in this study. It is the goal of the proposed study to compare the efficacy, as assessed primarily by sputum weight, of these two different devices (the Electroflo 500 and the G5 Flimm-Fighter) for airway clearance (AC) in CF patients with mild to moderate lung disease, who have stable lung health and perform AC at home as part of their routine therapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF established by standard criteria (sweat chloride > 60 mmol/L and/or two alleles affected by gene mutations know to be associated with CF).
2. Age older than 8 years.
3. Known to consistently produce sputum.
4. Currently on a home therapeutic regimen that includes some form of AC performed at least 1 time daily.
5. FEV1 > 30%-predicted, and with stable lung function

Exclusion Criteria:

1. Hospitalization for CF pulmonary complications in the 1 months preceding enrollment.
2. Hemoptysis > 60 cc in a single episode in the 4 weeks preceding enrollment.
3. Chronic chest pain.
4. Participation in another interventional clinical trial in the previous 30 days.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Milla, MD, Principal Investigator — Stanford University

RESULTS

PARTICIPANT FLOW:
Groups:
- Electro-Flo, Then G5: The patients were randomized to a series of airway clearance sessions with Electro-Flo on Day 1 and G5 on Day 2.
  Electro-Flo Intervention: An assigned respiratory therapist performed airway clearance on each participant with the Electro-Flo device following the 2012 CFF therapy guidelines
- G5, Then Electro-Flo: The patients were randomized to a series of airway clearance sessions with G5 on Day 1 and Electro-Flo on Day 2.
  G5 Intervention: An assigned respiratory therapist performed airway clearance on each participant with the G5 device following the 2012 CFF therapy guidelines
Period: Overall Study
Arm/Group | Electro-Flo, Then G5 | G5, Then Electro-Flo
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants had the diagnosis of cystic fibrosis. All enrolled had baseline sputum production and were deemed at their baseline health status.
Groups:
- All Study Participants: Electro-Flo Intervention: An assigned respiratory therapist performed airway clearance on each participant with the Electro-Flo device following the 2012 CFF therapy guidelines.
  G5 Intervention: An assigned respiratory therapist performed airway clearance on each participant with the G5 device following the 2012 CFF therapy guidelines.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 6
Basline Pulmonary Function (FEV1) [Mean (Standard Deviation); unit: Liters] | 2.42 (20.28)

OUTCOME MEASURES:

1. Primary Outcome: Wet Sputum Weight
Description: To compare the wet to dry weight of study patients' sputum collected during their Day 1 & Day 2 therapy sessions.
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: gram
Groups:
- ElectroFlo Arm: ElectroFlo Arm
- G5 Flimm Fighter Arm: G5 Flimm Fighter arm
Arm/Group | ElectroFlo Arm | G5 Flimm Fighter Arm
Number analyzed (Participants) | 25 | 25
gram | 5.22 [0 to 11.2] | 4.19 [0 to 8.56]

2. Secondary Outcome: Pulmonary Function Measured as a Percent Predicted BEFORE Therapy With Either ElectroFlo 5000 / G5.
Description: Comparison of pulmonary function by doing spirometry testing on study patients during their Day 1 & Day 2 therapy sessions. Will also compare the results based on the therapies they receive.
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: percentage of predicted value
Groups:
- Electro-Flo Arm: Electro-Flo arm
  Electro-Flo Intervention: An assigned respiratory therapist performed airway clearance on each participant with the Electro-Flo device following the 2012 CFF therapy guidelines
- G5 Arm: G5 arm
  G5 Intervention: An assigned respiratory therapist performed airway clearance on each participant with the G5 device following the 2012 CFF therapy guidelines
Arm/Group | Electro-Flo Arm | G5 Arm
Number analyzed (Participants) | 25 | 25
percentage of predicted value | 69.16 [49.25 to 89.07] | 69.84 [49.61 to 90.07]

3. Secondary Outcome: PRO (Patient-reported Outcome)
Description: Investigators will question the study patients re: their tolerability and comfort after the intervention on Day 1 & Day 2 visits.
Time Frame: End of study visit per intervention
Population: Patients rated comfort on a scale of 1 (most comfortable) to 10 (most un-comfortable)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Electro-Flo Arm | G5 Arm
Number analyzed (Participants) | 25 | 25
units on a scale | 3.24 [1.03 to 5.45] | 3.2 [0.58 to 5.82]

4. Primary Outcome: Dry Sputum Weight
Description: To compare the wet to dry weight of study patients' sputum collected during their Day 1 & Day 2 therapy sessions.
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: gram
Groups:
- Electro-Flo Arm: Electro-Flo arm Electro-Flo device following the 2012 CFF therapy guidelines
Arm/Group | Electro-Flo Arm | G5 Arm
Number analyzed (Participants) | 25 | 25
gram | 0.21 [0 to 0.54] | 0.15 [0 to 0.33]

5. Primary Outcome: Pulmonary Function Measured as a Percent Predicted AFTER Therapy With Either ElectroFlo 5000 / G5.
Description: as for outcome 2
Time Frame: End of study visit per intervention
Measure: Mean (Full Range); unit: percentage of predicted value
Arm/Group | Electro-Flo Arm | G5 Arm
Number analyzed (Participants) | 25 | 25
percentage of predicted value | 71.36 [51.08 to 91.64] | 71.52 [51.45 to 91.59]

ADVERSE EVENTS:
Groups:
- Electro Flo: Electro flo
- G5 Flimm Fighter: G5 Flimm Fighter
Arm/Group | Electro Flo | G5 Flimm Fighter
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes